CLINICAL TRIAL: NCT02576015
Title: The Effect of Continuous Femoral Nerve Block With Modulation of Depth of Anesthesia on Prognosis of Patients Receiving Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Min Su (Other)
Responsible Party: Sponsor-Investigator, Min Su, Chief of the Departmemt of Anesthesiology, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CYYYMZK-07
Record Dates: First submitted 2015-10-08; First posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Pain Management; Sedation; Peripheral Nerve Block; Total Knee Arthroplasty
MeSH Terms: conditions — Agnosia | interventions — Lidocaine; Ultrasonography; Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group L (Experimental): Participants in group L will receive a single injection for femoral nerve block combined with continuous femoral nerve block intra-operatively. The femoral nerve block will be performed before the induction of anesthesia on the leg to be operated. Then the patients were given the 2% lidocaine 10 ml and 1% ropivacaine 10 ml as initial dose,then,the patients will receive a continuous infusion of 0.15% ropivacaine at 15 ml/h.Intra-operatively, bispectral index score (BIS) was titrated with the adjusting of desflurane to maintain the index between 50-60.After the surgery,these patients will receive continuous femoral nerve analgesia till 3 days post-operatively( the loading dose was set at 5 ml of 0.15% ropivacaine followed by an infusion of 0.15% ropivacaine at 5 ml/h, with bolus of 5 ml and the lock time of 30 min).
  Interventions: Procedure: peri-operative continuous femoral nerve block with light sedation; Drug: lidocaine; Device: ultrasound; Device: insulated needle (Contiplex B Braun, Melsungen, Germany); Drug: ropivacaine
- Group D (Sham Comparator): Participants in group D will receive the placement of femoral nerve catheter preoperatively. The same dose of 0.9% saline was injected and infused as group L intra-operatively. Bispectral index score (BIS) was titrated with the adjusting of desflurane to maintain the index between 30-40.After the surgery,these patients will receive continuous femoral nerve analgesia till 3 days post-operatively( the loading dose was set at 5 ml of 0.15% ropivacaine followed by an infusion of 0.15% ropivacaine at 5 ml/h, with bolus of 5 ml and the lock time of 30 min).
  Interventions: Procedure: post-operative continuous femoral nerve block; Device: ultrasound; Drug: ropivacaine; Drug: saline

INTERVENTIONS:
Procedure: peri-operative continuous femoral nerve block with light sedation — this technique will be administered to participants in group L .The puncture site was identified using ultrasound guidance (2 cm distal to the inguinal ligament, and 1 ～2 cm lateral to the femoral artery).2% lidocaine was used for topical anesthesia, then an insulated needle (Contiplex B Braun, Melsungen, Germany) (20 G*45 mm，short bevel，30°) was connected to the nerve stimulator（Innervator，Fisher &Paykel，New Zealand）.The parameters were as follows: stimulating intensity of 1 mA at a rate of 2 Hz. The needle was advanced at 30°～45° angle to the skin, until quadriceps femoral muscle twitches were elicited. Its position was accepted if contractions were still elicited when an output equal to 0.3 mA.The participants will receive continuous femoral nerve block intra-operatively and post-operatively till 3 days post-operatively.The depth of anesthesia will modulated at 50-60 with BIS monitoring
  Arms: Group L
Procedure: post-operative continuous femoral nerve block — this technique will be administered to participants in group D .The puncture site was identified using ultrasound guidance (2 cm distal to the inguinal ligament, and 1 ～2 cm lateral to the femoral artery).2% lidocaine was used for topical anesthesia, then an insulated needle (Contiplex B Braun, Melsungen, Germany) (20 G*45 mm，short bevel，30°) was connected to the nerve stimulator（Innervator，Fisher &Paykel，New Zealand）.The parameters were as follows: stimulating intensity of 1 mA at a rate of 2 Hz. The needle was advanced at 30°～45° angle to the skin, until quadriceps femoral muscle twitches were elicited. Its position was accepted if contractions were still elicited when an output equal to 0.3 mA.The participants will receive continuous femoral nerve block post-operatively till 3 days post-operatively.The depth of anesthesia will modulated at 30-40 with BIS monitoring
  Arms: Group D
Drug: lidocaine
  Arms: Group L
Device: ultrasound
Device: insulated needle (Contiplex B Braun, Melsungen, Germany)
  Arms: Group L
Drug: ropivacaine
Drug: saline
  Arms: Group D

SUMMARY:
The interaction of analgesia and sedation ot their effect on the prognosis of surgical patients still need to be elucidated.Currently, how to optimize intra-operative Analgesia and sedation to improve the prognosis of surgical patients is still a mystery.Intra-operative nerve block provided regional analgesia of the operated knee, which reduced the dosages of sedatives and analgesics.Based on a pilot study,the investigators found a decrease of post-operative adverse composite outcomes with the use of continuous femoral nerve block (2% versus 7%) ,therefore, the investigators postulate that general analgesia with lighter sedation in combination with peripheral nerve block could reduce the post-operative morbidity compared with deeper sedation.This randomized controlled trial is designed to test this hypothesis in patients receiving unilateral knee arthroplasty.

DETAILED DESCRIPTION:
This study was approved by the institutional review board of the First Affiliated Hospital of Chongqing Medical University. The protocol design is in accordance with Consolidated Standards of Reporting Trials (CONSORT) statement.This study is designed as a randomized controlled trial to compare intra-operative continuous femoral nerve block combined with lighter anesthetic depth (group L) with deeper anesthetic depth (group D) monitored by bispectral index (BIS). All potentially eligible participants will be asked to give written informed consent before they are enrolled in this study.The following outcomes will be assessed:post-operative major complications (post-operative pulmonary infection,need of mechanical respiratory support,myocardio-infarction,deep venous thrombosis, pulmonary embolism, stroke, poor wound healing,all-cause post-operative death within 30 days).Secondary Outcomes included :acute post-operative pain assessed by visual analogue scale and dosages of rescue medications;Dosages of intra-operative vasopressors,anesthetics and analgesics;Life quality measured by EQ-5D questionnaire 3 months post-operatively;adverse events associated with the femoral catheter (displacement, infection, hematoma,drop-out of catheter).

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the 18 years and younger than 80 years old
* Scheduled to receive selective unilateral knee replacement.

Exclusion Criteria:

* Bilateral knee replacement
* The secondary knee revision and knee surgery not interfering with articular joint cavity (wound debridement and suture)
* American Society of Anesthesiology (ASA) classification of anesthesia risk IV and V grade
* Body mass index higher than 35
* Coagulation dysfunction, which is assessed by activated partial thromboplastin time (APTT) higher than the upper limit by 10s; prothrombin time (PT) higher than the upper limit by 5s; International Normalized Ratio (INR) higher than 1.3, or any of criteria met above;
* Pre-operative hypoxia (SpO2< 90% or PO2<60 mmHg)
* Pre-operative hypercapnia (PCO2> 50 mmHg)
* Local infection of puncture sites
* Neurological diseases and pre-operative psychological disorders
* Uncontrolled general infection
* Intra-operative cardiac arrest.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Major post-operative complications | From the end of surgery to 30 days post-operatively
  Major post-operative complications summed the incidence of major complications post-operatively( (post-operative pulmonary infection,need of mechanical respiratory support,myocardio-infarction,deep venous thrombosis, pulmonary embolism, stroke, poor wound healing,all-cause post-operative death within 30 days),participants with at least one episode of the complications will be calculated as participants with complications,both the number of participants and number of events will be calculated.

SECONDARY OUTCOMES:
Acute post-operative Pain assessed by visual analogue scale | At 12 hours ,24hours ,48hours,72 hours post-operatively
  Acute
Dosages of rescue medications (mg) | From the end of surgery to 3 days post-operatively
  the dosages of tramadol,pethidine and Parecoxib during the use of patient controlled analgesia (PCA) post-operatively
Dosages of intra-operative vasopressors,anesthetics and analgesics | during the surgery
Life quality measured by euro-quality-5 dimensions (EQ-5D) | 3 months post-operatively
  EQ-5D is a commonly used scale for calibration of life quality
Adverse events associated with the femoral catheter | From the insertion of the catheter to 3 days post-operatively
  local infection,hematoma,drop-out of the catheter,nerve injury

CONTACTS AND LOCATIONS:
Overall Officials: Su Min, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Department of Anesthesiology,the first Affiliated Hospital of Chongqing Medical University, Chonqqing, Chongqing Municipality, China

REFERENCES:
- [Background] Singelyn FJ, Deyaert M, Joris D, Pendeville E, Gouverneur JM. Effects of intravenous patient-controlled analgesia with morphine, continuous epidural analgesia, and continuous three-in-one block on postoperative pain and knee rehabilitation after unilateral total knee arthroplasty. Anesth Analg. 1998 Jul;87(1):88-92. doi: 10.1097/00000539-199807000-00019. PMID 9661552
- [Background] Lieberman JR, Freiberg AA, Lavernia CJ. Practice management strategies among members of the American Association of Hip and Knee Surgeons. J Arthroplasty. 2012 Sep;27(8 Suppl):17-9.e1-6. doi: 10.1016/j.arth.2012.02.030. Epub 2012 Apr 12. PMID 22503334
- [Background] Wegener JT, van Ooij B, van Dijk CN, Karayeva SA, Hollmann MW, Preckel B, Stevens MF. Long-term pain and functional disability after total knee arthroplasty with and without single-injection or continuous sciatic nerve block in addition to continuous femoral nerve block: a prospective, 1-year follow-up of a randomized controlled trial. Reg Anesth Pain Med. 2013 Jan-Feb;38(1):58-63. doi: 10.1097/AAP.0b013e318272523c. PMID 23104147
- [Background] Morin AM, Kratz CD, Eberhart LH, Dinges G, Heider E, Schwarz N, Eisenhardt G, Geldner G, Wulf H. Postoperative analgesia and functional recovery after total-knee replacement: comparison of a continuous posterior lumbar plexus (psoas compartment) block, a continuous femoral nerve block, and the combination of a continuous femoral and sciatic nerve block. Reg Anesth Pain Med. 2005 Sep-Oct;30(5):434-45. doi: 10.1016/j.rapm.2005.05.006. PMID 16135347
- [Background] Law CJ, Jacobson GM, Kluger M, Chaddock M, Scott M, Sleigh JW. Randomized controlled trial of the effect of depth of anaesthesia on postoperative pain. Br J Anaesth. 2014 Apr;112(4):675-80. doi: 10.1093/bja/aet419. Epub 2013 Dec 8. PMID 24322572
- [Background] Baldini G, Bagry H, Carli F. Depth of anesthesia with desflurane does not influence the endocrine-metabolic response to pelvic surgery. Acta Anaesthesiol Scand. 2008 Jan;52(1):99-105. doi: 10.1111/j.1399-6576.2007.01470.x. Epub 2007 Nov 1. PMID 17976225
- [Background] Soumpasis I, Kanakoudis F, Vretzakis G, Arnaoutoglou E, Stamatiou G, Iatrou C. Deep anaesthesia reduces postoperative analgesic requirements after major urological procedures. Eur J Anaesthesiol. 2010 Sep;27(9):801-6. doi: 10.1097/EJA.0b013e328337cbf4. PMID 20679774
- [Background] Sahni N, Anand LK, Gombar K, Gombar S. Effect of intraoperative depth of anesthesia on postoperative pain and analgesic requirement: A randomized prospective observer blinded study. J Anaesthesiol Clin Pharmacol. 2012 Apr;28(2):266-7. doi: 10.4103/0970-9185.94920. No abstract available. PMID 22557763
- [Background] Whitlock EL, Villafranca AJ, Lin N, Palanca BJ, Jacobsohn E, Finkel KJ, Zhang L, Burnside BA, Kaiser HA, Evers AS, Avidan MS. Relationship between bispectral index values and volatile anesthetic concentrations during the maintenance phase of anesthesia in the B-Unaware trial. Anesthesiology. 2011 Dec;115(6):1209-18. doi: 10.1097/ALN.0b013e3182395dcb. PMID 22037642
- [Background] Kertai MD, Palanca BJ, Pal N, Burnside BA, Zhang L, Sadiq F, Finkel KJ, Avidan MS; B-Unaware Study Group. Bispectral index monitoring, duration of bispectral index below 45, patient risk factors, and intermediate-term mortality after noncardiac surgery in the B-Unaware Trial. Anesthesiology. 2011 Mar;114(3):545-56. doi: 10.1097/ALN.0b013e31820c2b57. PMID 21293252
- [Background] Leslie K, Myles PS, Forbes A, Chan MT. The effect of bispectral index monitoring on long-term survival in the B-aware trial. Anesth Analg. 2010 Mar 1;110(3):816-22. doi: 10.1213/ANE.0b013e3181c3bfb2. Epub 2009 Nov 12. PMID 19910621
- [Background] Punjasawadwong Y, Boonjeungmonkol N, Phongchiewboon A. Bispectral index for improving anaesthetic delivery and postoperative recovery. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD003843. doi: 10.1002/14651858.CD003843.pub2. PMID 17943802
- [Background] Willingham MD, Karren E, Shanks AM, O'Connor MF, Jacobsohn E, Kheterpal S, Avidan MS. Concurrence of Intraoperative Hypotension, Low Minimum Alveolar Concentration, and Low Bispectral Index Is Associated with Postoperative Death. Anesthesiology. 2015 Oct;123(4):775-85. doi: 10.1097/ALN.0000000000000822. PMID 26267244
- [Background] Gurman GM, Popescu M, Weksler N, Steiner O, Avinoah E, Porath A. Influence of the cortical electrical activity level during general anaesthesia on the severity of immediate postoperative pain in the morbidly obese. Acta Anaesthesiol Scand. 2003 Aug;47(7):804-8. doi: 10.1034/j.1399-6576.2003.00148.x. PMID 12859299
- [Background] Peng J, Wang SD. Effect of anesthesia combined with intercostal nerve block on analgesia for esophageal cancer after operation. Eur Rev Med Pharmacol Sci. 2015 Jun;19(12):2293-6. PMID 26166657
- [Background] Kratz T, Dette F, Schmitt J, Wiesmann T, Wulf H, Zoremba M. Impact of regional femoral nerve block during general anesthesia for hip arthoplasty on blood pressure, heart rate and pain control: A randomized controlled study. Technol Health Care. 2015;23(3):313-22. doi: 10.3233/THC-150898. PMID 25669214
- [Background] De Baerdemaeker LE, Struys MM, Jacobs S, Den Blauwen NM, Bossuyt GR, Pattyn P, Mortier EP. Optimization of desflurane administration in morbidly obese patients: a comparison with sevoflurane using an 'inhalation bolus' technique. Br J Anaesth. 2003 Nov;91(5):638-50. doi: 10.1093/bja/aeg236. PMID 14570784
- See also: CONsolidated Standards of Reporting Trials he Consort Group aimed at transparent reporting of the trial," — http://www.consort-statement.org